CLINICAL TRIAL: NCT04483440
Title: Phase 1 Open-Label, Dose-Escalation Study of the Safety, Tolerability and Preliminary Efficacy of Intravitreal 4D-110 in Patients With Choroideremia
Brief Title: Dose Escalation Study of Intravitreal 4D-110 in Patients With Choroideremia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: 4D Molecular Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4D-110-CP-0001
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Choroideremia
Keywords: CHM; transgene; gene therapy; AAV
MeSH Terms: conditions — Choroideremia

STUDY DESIGN:
Intervention Model Description: Each dose escalation cohort will initially recruit up to 3 patients to receive a single uniocular intravitreal injection of 4D-110 in a standard 3+3 design. The cohort will be expanded in the event of a dose limiting toxicity (DLT). Once the maximum tolerated dose (MTD)/maximum feasible dose (MFD) has been identified, up to 4 additional patients may be enrolled at that dose level to provide additional safety information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 4D-110 Dose 1 (Experimental): 4D-110 IVT injection
  Interventions: Biological: 4D-110
- 4D-110 Dose 2 (Experimental): 4D-110 IVT injection
  Interventions: Biological: 4D-110
- 4D-110 Dose 3 (Experimental): 4D-110 IVT injection
  Interventions: Biological: 4D-110

INTERVENTIONS:
Biological: 4D-110 — 4D-110 drug product developed for gene therapy which comprises an AAV capsid variant (4D-R100) carrying a transgene encoding a codon-optimized human CHM gene.

SUMMARY:
This study will evaluate safety, tolerability, and preliminary efficacy of a single intravitreal (IVT) injection of a recombinant adeno-associated virus (AAV) gene therapy, 4D-110, in male patients with genetically-confirmed Choroideremia (CHM).

DETAILED DESCRIPTION:
This is an open-label, Phase 1 study to evaluate safety and tolerability as well as preliminary efficacy of a single IVT injection of 4D-110 at three dose levels in male patients with genetically-confirmed CHM.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of CHM defined as a pathogenic mutation in the CHM gene, confirmed by genetic testing
* Both eyes must have ≥ 34 ETDRS letters (~20/200)

Key Exclusion Criteria:

* Clinically significant, active ocular or peri-ocular infection or inflammation in the study eye
* Patient has previously received any AAV treatment
* Ocular conditions or ocular media opacity in either eye that would preclude the planned treatment (i.e. IVT injection) or interfere with the interpretation of study endpoints (e.g. significant lens opacity)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2027-05-26 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of ocular and systemic adverse events (AEs) | 24 months
  Frequency and severity of ocular and systemic AEs including clinically significant changes in ocular evaluations, systemic examinations and laboratory testing.

CONTACTS AND LOCATIONS:
Overall Officials: Schonmei Lee, MD, Study Director — 4D Molecular Therapeutics
Locations (2):
- United States (2):
  - Retina Foundation of the Southwest, Dallas, Texas
  - Moran Eye Center, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No